CLINICAL TRIAL: NCT04700540
Title: A Mobile Informatics Solution to Aid in Memory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Advanced Medical Electronics (Other); University of Michigan (Other); Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SPH-2023-31117
Record Dates: First submitted 2020-12-17; First posted 2021-01-08 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease; Dementia
Keywords: Dementia; Alzheimer Disease; Social Interaction; Quality of Life
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: Researchers will enroll 100 PWMC and their care partners to participate in initial, 3-month, and 6-month surveys. Half of the PWMCs will be randomly assigned to the intervention group (to receive the SR) and the other half randomly assigned to the attention control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The PWMC and Care partner in this group will receive the SR. The project will provide a smartwatch and smartphone for the dyads in the study. All others (family, friends, etc.) will be able to download a smartphone app from an online store. Instructional material will be created to show the suggested information that can be entered into the app. Care partners and PWMC are administered surveys at baseline and 3 months following enrollment.
  Interventions: Device: Smartwatch Reminder (SR) system
- Attention Control Group (No Intervention): Care partners are administered surveys at baseline and 3 months following enrollment. The attention control group will receive a contact call from one of the researchers 3-months after enrollment. Based on our prior experience, PWMC and care partners in an attention control group will often seek information and psychosocial support during these calls. We will provide free information resources (e.g., brochures or websites of the Alzheimer's Association) at that time.

INTERVENTIONS:
Device: Smartwatch Reminder (SR) system — The Smartwatch Reminder (SR) system will automatically transmit pictures and relevant information, such as name or relationship, to a smartwatch worn by the PWMC when family or friends visit.
  Arms: Intervention Group

SUMMARY:
The researchers propose to develop an informatics system to assist people with memory impairment. Persons with Memory Concern (PWMC) recognize the faces they see daily, such as a spouse or caregiver, but they may confuse visiting friends and grandchildren or they may not match names with faces well. The inability to remember names or relationships contributes to isolation and deeply affects their social lives. The proposed solution is a Smartwatch Reminder (SR) system to conspicuously provide this information to the PWMC when needed. The system will be evaluated on the target persons with memory concern population to measure engagement and improvements in social interactions and quality of life.

DETAILED DESCRIPTION:
This research will evaluate technology designed to improve the quality of life for persons with dementia through external aids to assist with remembering. The primary goal of the Smartwatch Reminder (SR) is to facilitate social interaction for Persons with Memory Concern (PWMC) by providing facial recognition of family, friends, and other key people. The SR will be evaluated using an embedded experimental mixed methods design that combines the collection and analysis of qualitative data within a traditional randomized controlled trial design. To do so, researchers will enroll 100 PWMC and their care partners to participate in initial, 3-month, and 6-month surveys. Half of the PWMCs will be randomly assigned to the intervention group (i.e. receive the SR) and the other half randomly assigned to the attention control group. Each participant will take part in the study for a total of 6 months. All study procedures and data analysis are anticipated to be completed within 24 months.

ELIGIBILITY:
Inclusion criteria for PWMC are as follows:

* English speaking
* a physician diagnosis of early-stage Alzheimer's disease or mild-to-moderate cognitive impairment
* no history of serious mental illness (i.e., any major psychiatric disorder)

Inclusion criteria for care partners of PWMC are as follows:

* English speaking
* 21 years of age or over
* self-identifies as someone who provides assistance to the PWMC because of their memory loss (these individuals are called ''care partners,'' as these individuals may or may not provide the intensive hands-on care typical of ''caregivers'')
* plans to remain in the area for at least 6 months in order to reduce loss to follow-up
* indicates a willingness to use the smartwatch system

Exclusion Criteria for PWMC are as follows:

* non-English speaking
* no physician diagnosis of early-stage Alzheimer's disease or mild-to-moderate cognitive impairment
* a history of serious mental illness (i.e., any major psychiatric disorder)

Exclusion criteria for care partners of PWMC are as follows:

* non-English speaking
* under 21 years of age
* does not identify as someone who provides assistance to the PWMC because of their memory loss
* does not plan on remaining in the area for at least 6 months
* does not indicate a willingness to use the smartwatch system

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Public access to the research data generated from this project will be offered via de-identified data files maintained by the investigators. All personal identifiers of family caregivers of persons with Alzheimer's disease or a related dementia (ADRD) participating in the study will be removed and replaced with random identification numbers prior to distributing data files. Potential external investigators will be asked to complete a data use agreement and a recommended citation to these materials will be provided. Data from the project will be maintained on a secure University of Minnesota School of Public Health shared server for 3 years following study completion.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 81 caregivers consented and 81 persons with memory concerns consented or assented to be part of the study, totaling 162 participants or 81 dyads. Six participants or 3 dyads withdrew before randomization. Data is reported for the 156 randomized participants.
Groups:
- Intervention Group: The PWMC and Care partner in this group will receive the SR. The project will provide a smartwatch and smartphone for the dyads in the study. All others (family, friends, etc.) will be able to download a smartphone app from an online store. Instructional material will be created to show the suggested information that can be entered into the app. Care partners and PWMC are administered surveys at baseline, 3 months and 6 months following enrollment.
  Smartwatch Reminder (SR) system: The Smartwatch Reminder (SR) system will automatically transmit pictures and relevant information, such as name or relationship, to a smartwatch worn by the PWMC when family or friends visit.
- Attention Control Group: Care partners are administered surveys at baseline, 3 months and 6 months following enrollment. The attention control group will receive a contact call from one of the researchers 3-months and 6-months after enrollment. Based on our prior experience, PWMC and care partners in an attention control group will often seek information and psychosocial support during these calls. We will provide free information resources (e.g., brochures or websites of the Alzheimer's Association) at that time.
Period: Overall Study
Arm/Group | Intervention Group | Attention Control Group
Started | 84 (84 individual participants, 42 dyads were part of the intervention group.) | 72 (72 individual participants or 36 dyads were part of the control group)
Completed | 44 (44 individual participants or 22 dyads completed the intervention group) | 64 (64 individual participants or 32 dyads finished in the the control group)
Not Completed | 40 | 8
Not completed — Withdrawal by Subject | 12 | 8
Not completed — Participant wished to discontinue intervention use, but remained in study to complete surveys only. | 28 | 0

BASELINE CHARACTERISTICS:
Population: While 162 individuals (81 dyads) initially enrolled in the study, only 156 individuals (78 dyads) completed the baseline survey and moved to randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Attention Control Group | Total
Number analyzed (Participants) | 84 | 72 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (13.3) | 69.8 (10.7) | 69.9 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 46 | 98
  Male | 32 | 26 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 80 | 66 | 146
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 3 | 1 | 4
  White | 70 | 64 | 134
  More than one race | 4 | 4 | 8
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: PWMC Loneliness
Description: Original three-item measure, including:
  * How often do you feel you lack companionship?
  * How often do you feel left out?
  * How often do you feel isolated from others? Scale range 3-9, higher scores indicate higher rates of social isolation.
Time Frame: 3 months
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Group | Attention Control Group
Number analyzed (Participants) | 28 | 31
units on a scale | 4.90 [4.23 to 5.13] | 5.28 [4.63 to 5.53]

2. Primary Outcome: PWMC Social Relationships and Social Support
Description: The Lubben Social Network Scale (LSNS) is a measure of social relationships and social support networks. We used the shortened 6-item scale to reduce test burden. The 6-item scale has a range of 0 - 30 with higher scores indicating more robust social networks / access to support.
Time Frame: 3 months
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Intervention Group | Attention Control Group
Number analyzed (Participants) | 28 | 31
units on a scale | 13.50 [11.70 to 15.3] | 10.72 [8.92 to 12.52]

3. Secondary Outcome: PWMC Physical and Mental Well-being
Description: We used the Global Health Scale. This tool is designed to assess an individual's overall physical and mental wellbeing. The scale measures subjective health perceptions. Scale scores range from 0 - 100, with higher scores indicating higher rates of mental and physical well-being.
Time Frame: 3 months
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group | Attention Control Group
Number analyzed (Participants) | 28 | 31
score on a scale | 32.69 [26.68 to 38.70] | 32.72 [26.71 to 38.73]

ADVERSE EVENTS:
Time Frame: Adverse events were documented during study enrollment (following consent through final data collection). Participants were enrolled for about 6 months.
Arm/Group | Intervention Group | Attention Control Group
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/72
Serious Adverse Events (participants affected / at risk) | 1/84 | 2/72
Other Adverse Events (participants affected / at risk) | 5/84 | 5/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Group (N=84) | Attention Control Group (N=72)
Person with Memory Concerns Stroke (Cardiac disorders) | 1 | 1 — Caregiver shared the person with memory concerns experienced a stroke.
Suicidal Ideation (Psychiatric disorders) | 0 | 1 — Caregiver indicated that the person with memory concerns had been hospitalized for suicidal ideation due to medication side effects
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Group (N=84) | Attention Control Group (N=72)
Diabetes hospitalization (Vascular disorders) | 1 | 0
PWMC Fractured Pelvis (Injury, poisoning and procedural complications) | 1 | 0 — Person with memory concerns fractured their pelvis.
Weather related fall (Injury, poisoning and procedural complications) | 1 | 0 — Caregiver fell on ice resulting in surgery.
Low blood pressure (Cardiac disorders) | 1 | 0 — Caregiver shared that a change in their regular activity was due to low blood pressure.
Eye Surgery (Eye disorders) | 1 | 0 — Caregiver shared that the person with memory concerns had eye surgery.
Knee replacement (Musculoskeletal and connective tissue disorders) | 0 | 1 — Care giver had a planned knee replacement surgery.
Back surgery (Musculoskeletal and connective tissue disorders) | 0 | 1 — Caregiver had planned back surgery
PWMC Instability and memory concerns (Congenital, familial and genetic disorders) | 0 | 1 — CG shared that the PWMC was needing more outpatient doctor visits for instability and memory concerns.
Person with memory concerns flu (Infections and infestations) | 0 | 1 — Caregiver shared the PWMC had flu weeks earlier.
Sepsis (Blood and lymphatic system disorders) | 0 | 1 — Caregiver hospitalized for sepsis due to kidney infection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/40/NCT04700540/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/40/NCT04700540/ICF_001.pdf